CLINICAL TRIAL: NCT05159206
Title: Evaluation of a Novel CT-based 3D Planning, Computer Navigation and Subsequent Migration Analysis in Total Hip Arthroplasty: A Single Arm Study With 2 Years Follow-up
Brief Title: CT-based 3D Planning, Computer Navigation and Subsequent Migration Analysis in Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTS plan, nav, migr
Record Dates: First submitted 2021-10-26; First posted 2021-12-16 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Hip Osteoarthritis
Keywords: Hip Osteoarthritis; Total Hip Arthroplasty; CT templating; CT migration analysis; CT navigation
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: One group of patients undergoing total hip arthroplasty with a new technique of preoperative templating, per-operative navigation and postoperative migration analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CT group (Other): CT-scan preoperatively, postoperatively and at 3 months, 1 and 2 years. Per-operative navigation based on the CT scan.
  Interventions: Procedure: CT group

INTERVENTIONS:
Procedure: CT group — This group will do a preoperative CT scan for templating. The same scan is then used for per-operative navigation. After surgery, a postoperative CT will validate the templating/navigation, and then subsequent CT scans (postoperative, 3 months, 1 and 2 years) will be done to measure prosthetic migration over time.
  Other Names: RSA-follow up; CT-based Navigation

SUMMARY:
The aim of this study is to evaluate a new technique that optimizes the prosthesis position for patients who undergo total hip arthroplasty surgery. Today, most surgeons take a regular X-ray (2D) to plan the surgery. In this study, patients will do a computed tomography (CT) before surgery, and with the use of the new system, the investigators will be able to make a more accurate plan when it comes to prosthetic placement and leg length adjustment in 3D. The software uses artificial intelligence (AI) to generate the information required for clinical conclusions automatically, and it enables surgeons to adapt to each unique case and anticipate situations during surgery. The system also helps the surgeon during operation with a navigation tool to place the implant in the pre-operatively planned position. It guides surgeons in real-time to place the implants accurately. To see whether the plan and navigation were correct, the investigators will do a new computed tomography after surgery to look at the achieved result.

In addition to planning and navigation, the same system can be used to measure the migration of the prosthesis in relation to the bone over time using AI by comparing multiple scans. The investigators aim to follow all patients for 2 years (total of 4 CT scans after surgery) with the intention to be able to foresee implant loosening.

DETAILED DESCRIPTION:
The aim of this study is to evaluate a new system for CT-based 3D planning, navigation and subsequent postoperative migration analysis in patients with total hip arthroplasty (THA). Patients (age 40-75 years) with osteoarthritis, eligible for surgery, are asked to participate, and the investigators plan to follow all patients for 2 years after surgery.

In THA surgery, the goal is to recreate the natural motion-center of the hip, adjust for possible leg length differences and to optimize prosthetic placement to reduce the risk of future dislocation or loosening. Today, usually a plain X-ray is taken before the operation to plan size and position. This has its limitations since the surgeon can not assess the 3D position on a 2D image. In this study, the investigators are using a new system for planning in 3D, based on a low-dose CT scan and with the help of AI. Moreover, the surgeon get real-time information of the prosthetic position during surgery (called navigation), after matching the physical patient to a virtual patient. The hypothesis is that prosthetic placement and patient satisfaction will improve with 3D planning and navigation, resulting in a more anatomical restoration, and that postoperative complications, such as dislocation and ultimately loosening will reduce.

Entering this study entails taking a CT scan before surgery (instead of a plain X-ray), and for validation, a postoperative CT scan. This enables the investigators to find out whether the planning and navigation are confirmed by the postoperative position. In addition to planning and navigation, the investigators wish to implement a way of measuring prosthetic migration after surgery. Today, this is done by implanting small metal (tantalum) markers in the bone during surgery, and then measuring the distance between prosthesis and markers over time in a special software on multiple X-rays (This method is called RSA, Radiostereometric Analysis). However, few hospitals have the expertise or equipment to do these analyses and it is a somewhat laborious process. This study will evaluate a new tool for making equivalent migration analysis, based on CT scans. By matching the postoperative CT image to subsequent CT scans at 3 months, 1 and 2 years after surgery, the investigators can see how much the prosthesis has moved in relation to the bone and hopefully being able to foresee future loosening. The hypotheses is that CT migration analysis will be as accurate and precise as the current gold standard (RSA). A subset of the patients will have RSA performed as well for direct comparison between the systems regarding migration.

A transition from plain X-ray images to low-dose CT will result in a marginal increase in the radiation dose. At the same time, it means that a much more accurate imaging of the skeleton is performed, and thus improved preoperative planning and a per-operative navigation can be done with much more predictable results. This study has been approved by the Swedish Ethical Review Authority, as well as the local radiation committee. The company, Ortoma, supplying the measurement system for planning and navigation (Ortoma Treatment Solution (OTS™)) has received ISO13485 certification and CE-certificate on all parts.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary hip osteoarthritis
* Qualified for total hip arthroplasty surgery at the regional Hospital

Exclusion Criteria:

* BMI >35
* Unable to comprehend the patient information
* Other cause for assessing the patient as ineligible (such as: serious medical comorbidity or active drug abuse)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
CT validation | Up to 10 days after surgery
  To validate the Ortoma treatment solution software, the investigators will compare the preoperative CT plan (planned prosthesis size and position) to the actual achieved postoperative implant size and position as measured on postoperative CT. The investigators will also compare the per-operatively measured values during surgical navigation to the measured values on postoperative CT. The measurements include translational (mm) and rotational (degrees) differences between planned, per-operative and achieved implant position, as well as offset and leg length differences (mm).
Change in prosthetic migration | First evaluation after 1 year and planned further at 2 years after surgery
  To measure migration over time (cup to pelvic bone and stem to femur bone) subsequent CT scans will be taken postoperative, at 3 months, 1 and 2 years after surgery. A subgroup of 10 patients will have RSA-follow up as well, at the same time intervalls, to compare to. The investigators will measure translational and rotational migration and if possible a 3D-vector.

SECONDARY OUTCOMES:
Forgotten Joint Score (FJS) | Up to 2 years after surgery (preop, 3 months, 1 and 2 years)
  Patients will be asked to fill in this patient reported outcome measure form (FJS) before, and after surgery
Hip dysfunction and Osteoarthritis Outcome Score (HOOS) | Up to 2 years after surgery (preop, 3 months, 1 and 2 years)
  Patients will be asked to fill in this patient reported outcome measure form (HOOS) before, and after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Flivik, MD PhD, Principal Investigator — Dept of Orthpaedics, Skane University Hospital, Sweden
Locations (1):
- Department of Orthopedics, Skåne University Hospital, Lund University, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
After study publication, IPD underlying the results will be available on reasonable request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication
Access Criteria: On reasonable request to the study investigators